CLINICAL TRIAL: NCT01464112
Title: A Phase 1b Dose Escalation Study of the Histone Deacetylase Inhibitor (HDACi) JNJ-26481585 in Combination With VELCADE (Bortezomib) and Dexamethasone for Subjects With Relapsed Multiple Myeloma
Brief Title: A Dose Escalation Study of the Histone Deacetylase Inhibitor (HDACi) JNJ 26481585 in Combination With VELCADE (Bortezomib) and Dexamethasone for Patients With Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018661; 26481585MMY1001 (Other: Janssen Research & Development, LLC); 2011-001001-27 (EudraCT Number)
Record Dates: First submitted 2011-08-30; First posted 2011-11-03 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma that has relapsed or is progressive following prior therapy; Relapsed Multiple Myeloma; JNJ 26481585; VELCADE; Bortezomib; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- 001 (Experimental)
  Interventions: Drug: JNJ-2641585 / VELCADE / Dexamethasone

INTERVENTIONS:
Drug: JNJ-2641585 / VELCADE / Dexamethasone — JNJ-26481585: type=range, unit=mg, number=6 to 12, form=capsules, route=oral use, on Days 1, 3, and 5 of each week. VELCADE: type=exact, unit=mg/m2, number=1.3, form=powder for solution for injection, route=subcutaneous use, on Days 1, 4, 8, and 11 of each 21-day cycle (Cycles 1 to 8) and on Days 1, 8, 15, and 22 of each 35-day cycle (Cycles 9-11). Dexamethasone: type=exact, unit=mg, number=20, form=tablets, route=oral use, on the day of and after VELCADE.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability and to establish the maximum tolerated dose of JNJ-26481585 combined with VELCADE and dexamethasone.

DETAILED DESCRIPTION:
This is an open-label (patient and study personnel will know what treatment is being administered), multicenter, dose escalation study. Increasing doses of JNJ-26481585 will be explored in combination with the standard VELCADE/dexamethasone dose. After the maximum tolerated dose (MTD) is determined, up to 24 patients will be entered in a treatment group to receive the MTD (and if deemed necessary a lower dose level) to further assess the safety and activity of this combination. There will be 3 phases in the study: a Screening Phase (from signing of informed consent until immediately before dosing), an open-label Treatment Phase (from the first dose of JNJ-26481585 and VELCADE-dexamethasone until the End of Treatment Visit), and a Posttreatment/Follow-up Phase. Patients who achieve a positive response to treatment at the end of Cycle 1 will continue to receive JNJ-26481585 and VELCADE-dexamethasone for a maximum of 11 cycles (eight 3-week treatment cycles, followed by three 5-week treatment cycles). Patients with progressive disease (PD) or unacceptable toxicity will be withdrawn from treatment. In the Follow-Up Phase, patients whose disease has not progressed or who discontinued treatment for reasons other than PD will be assessed approximately every 6 weeks until PD is recorded or until the start of subsequent therapy. The study will end when all patients have been assessed with PD, or 12 months after the last patient is enrolled, whichever is earlier. Patient safety will be monitored. Drug A, JNJ-26481585, will be taken orally on Days 1, 3, and 5 of each week at doses starting at 6 mg and escalating to 12 mg. Drug B, VELCADE, will be given by subcutaneous injection (under the skin) at a dose of 1.3 mg/m2 on Days 1, 4, 8, and 11 of each 21-day cycle (Cycles 1 to 8) and on Days 1, 8, 15, and 22 of each 35-day cycle (Cycles 9-11). Drug C, dexamethasone, will be taken orally on the day of and after VELCADE at a dose of 20 mg. Dosing may be adjusted, based on tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance status score 0-2
* Measurable or secretory multiple myeloma
* Relapse or progression of myeloma following prior systemic antineoplastic therapy
* Pretreatment clinical laboratory values meeting protocol-specified criteria
* Left ventricular ejection fraction rate within normal limits

Exclusion Criteria:

* Peripheral neuropathy or neuralgia >=2, according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0
* Diagnosis of primary amyloidosis, plasma cell leukemia, or other similar conditions
* Diagnosis of Waldenstrom macroglobulinemia with protocol-specified immunoglobulin levels
* Prior histone-deacetylase inhibitor therapy - More than 3 prior lines of therapy
* Cardiac risk factors: unstable angina or myocardial infarction within the preceding 12 months, congestive heart failure (New York Heart Association Class II-IV), known presence of dilated, hypertrophic, or restrictive cardiomyopathy
* Any other cardiac abnormality that, in the opinion of the investigator, medical monitor, or consultant cardiologist, may place the patient at an unacceptably increased risk with study drug
* History of any of the following: sustained ventricular tachycardia, ventricular fibrillation, Torsades de Pointes, atrial fibrillation, cardiac arrest, Mobitz II second degree heart block, or third degree heart block - QTc at Screening > 450 ms in males / > 470 ms in females
* Family history of short QT syndrome, long QT syndrome
* Obligate use of a cardiac pacemaker - Use of medications that may cause Torsades de Pointes

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09-16 (Actual); Primary Completion 2013-11-19 (Actual); Study Completion 2013-11-19 (Actual)

PRIMARY OUTCOMES:
Determine the dose-limiting toxicity and set the MTD for the combination of JNJ-26481585 and VELCADE-dexamethasone | Maximum of 18 months
  Based on the safety analysis of all cohorts using the patients-treated population

SECONDARY OUTCOMES:
Adverse events | Maximum of 18 months
  As a measure of safety
Clinical laboratory tests | Maximum of 18 months
  As a measure of safety
Overall response rate | Maximum of 18 months
Duration of response | Maximum of 18 months
Profile of pharmacokinetics evaluations for JNJ-26481585 | Maximum of 18 months
  Cmax, Area Under Curve, Tmax
Profile of pharmacokinetics evaluations for VELCADE | Maximum of 18 months
  Cmax, Area Under Curve, Tmax
Bone cell morphology | Maximum of 18 months
Pulse | Maximum of 18 months
Heart rate | Maximum of 18 months
Blood pressure | Maximum of 18 months
Body temperature | Maximum of 18 months
Height | Maximum of 18 months
Weight | Maximum of 18 months
Body surface area | Maximum of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC & Development, L.L.C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- France (3):
  - Lille
  - Nantes
  - Tours

REFERENCES:
- [Result] Moreau P, Facon T, Touzeau C, Benboubker L, Delain M, Badamo-Dotzis J, Phelps C, Doty C, Smit H, Fourneau N, Forslund A, Hellemans P, Leleu X. Quisinostat, bortezomib, and dexamethasone combination therapy for relapsed multiple myeloma. Leuk Lymphoma. 2016 Jul;57(7):1546-59. doi: 10.3109/10428194.2015.1117611. Epub 2016 Jan 12. PMID 26758913